CLINICAL TRIAL: NCT00883220
Title: Self-management of Urine Flow in Long-term Urinary Catheter Users
Brief Title: Self Management in Urinary Catheter Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Visiting Nurse Service of New York (Other)
Responsible Party: Principal Investigator, Mary Wilde, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01NR010553-01 (NIH); 1R01NR010553-01 (NIH)
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2011-07

CONDITIONS: Urinary Retention; Neurogenic Bladder
Keywords: self management; chronic condition; urinary catheter
MeSH Terms: conditions — Urinary Retention; Urinary Bladder, Neurogenic; Chronic Disease | interventions — Self-Management; Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-management of urinary catheter (Experimental): Intervention: Self-management group--teaching behavioral approaches(awareness, self-monitoring, and self-management) to prevent or minimize urinary catheter complications.
  Interventions: Behavioral: Self-management of urinary catheter
- Usual care 2 (No Intervention): Usual care for urinary catheter. Home care and/or clinic care is the usual care for people with long-term urinary catheters.

INTERVENTIONS:
Behavioral: Self-management of urinary catheter — Awareness, self-monitoring, and self-management of urine flow are taught. Focus is on attaining adequate and consistent levels of fluid intake and preventing catheter dislodgement.
  Other Names: self-management; self-monitoring; urinary catheter self care
  Arms: Self-management of urinary catheter

SUMMARY:
Learning to self-manage urine flow may help people prevent or minimize persistent complications from long-term indwelling urethral or suprapubic catheters.

DETAILED DESCRIPTION:
Urinary catheter users commonly experience adverse health effects, such as urinary tract infection (UTI), blockage, dislodgement, and leakage, leading to poor quality of life indicators. Catheter-related problems often require health care utilization resulting in increased health care costs. Self-management of urine flow is an essential part of self-care for people with long-term urinary catheters and may lead to prevention or reduction of catheter-related problems and improved quality of life.This study tests the effectiveness of a urinary catheter self-management intervention in a randomized trial of 220 patients, with 12 months of follow-up. The experimental intervention is designed to enhance self-management of urine flow in individuals with long-term urinary catheters, with the goal of decreasing catheter related complications and enhancing quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Have an indwelling urethral or suprapubic catheter and expect to use it for at least one year.
* Live in Central or Western New York State (Utica to Buffalo regions approximately)OR are cared for by the Visiting Nurse Service of New York City.
* Able to complete study measurements alone or with the help of a family member or caregiver.
* Able to communicate with the study personnel in English.
* Have access to a telephone for data collection.

Exclusion Criteria:

* Terminally ill
* Cognitively impaired
* No catheter associated UTI within the previous 12 months NOR blockage NOR dislodgement in the previous 6 months(only in people who have had the catheter for 12 months or more)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Symptomatic urinary tract infection | every two months for 12 months

SECONDARY OUTCOMES:
Urinary catheter quality of life | 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary H. Wilde, RN, PhD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Center for Home Care Policy & Research, Visiting Nurse Service of New York, New York, New York
  - Urinary of Rochester, Rochester, New York

REFERENCES:
- [Derived] Wilde MH, Crean HF, McMahon JM, McDonald MV, Tang W, Brasch J, Fairbanks E, Shah S, Zhang F. Testing a Model of Self-Management of Fluid Intake in Community-Residing Long-term Indwelling Urinary Catheter Users. Nurs Res. 2016 Mar-Apr;65(2):97-106. doi: 10.1097/NNR.0000000000000140. PMID 26938358
- [Derived] Wilde MH, McMahon JM, McDonald MV, Tang W, Wang W, Brasch J, Fairbanks E, Shah S, Zhang F, Chen DG. Self-management intervention for long-term indwelling urinary catheter users: randomized clinical trial. Nurs Res. 2015 Jan-Feb;64(1):24-34. doi: 10.1097/NNR.0000000000000071. PMID 25502058